CLINICAL TRIAL: NCT00976612
Title: Pharmacokinetic Study of Nilotinib in Patients With Metastatic or Unresectable Gastrointestinal Stromal Tumor Showing Failure to Both Imatinib and Sunitinib
Brief Title: Nilotinib Pharmacokinetics (PK) in Gastrointestinal Stromal Tumor (GIST): Nilotinib PK
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Other Study IDs: AMC0901
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal stromal tumor; pharmacokinetics; nilotinib
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — nilotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood about 4ml
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nilotinib: Patients who receive nilotinib with failure to both imatinib and sunitinib
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib 400mg bid daily

SUMMARY:
In patients who are receiving nilotinib, nilotinib plasma levels will be measured after 1 month of nilotinib treatment. The relationship between surgery type and nilotinib pharmakokinetic properties will be investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic or unresectable gastrointestinal stromal tumor
* Patients receiving nilotinib after failure to imatinib and sunitinib

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with metastatic or unresectable gastrointestinal stromal tumor who failed to imatinib and sunitinib.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2009-01; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
nilotinib pharmacokinetics | Up to 3years

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, M.D., PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea